CLINICAL TRIAL: NCT05170230
Title: The Effect of Intracapsular Injection of Terlipressin Versus Carbitocin on Hemoglobin and Blood Loss During Laparoscopic Myomectomy Operations: Double Blinded Randomized Placebo-Controlled Trial
Brief Title: The Effect of Intracapsular Injection of Terlipressin Versus Carbitocin on Hemoglobin and Blood Loss During Laparoscopic Myomectomy Operations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Elbanna Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Elbanna_006
Record Dates: First submitted 2021-12-06; First posted 2021-12-27 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-10

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — Terlipressin

STUDY DESIGN:
Intervention Model Description: This study is a prospective, comparative, double-blinded randomized placebo-controlled trial and multi-center study that will be conducted at Wael ElBanna Clinic and the NRC site
  The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms:
  * Arm 1: intracapsular myomectomy Terlipressin injection in women undergoing laparoscopic myomectomy procedure
  * Arm 2: intracapsular myomectomy Carbetocin injection in women undergoing laparoscopic myomectomy procedure
  * Arm 3: intracapsular myomectomy saline injection in women undergoing laparoscopic myomectomy procedure Subjects who meet diagnostic requirements as listed in the inclusion and exclusion criteria will be included in the study. Women will be randomized to one of the three arms using a computer-generated randomization table with a 1:1:1 group allocation.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intracapsular myomectomy Terlipressin injection (Active Comparator): intracapsular myomectomy Terlipressin injection in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin
- intracapsular myomectomy Carbetocin injection (Active Comparator): intracapsular myomectomy Carbetocin injection in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin
- intramyometrial saline (Placebo Comparator): intracapsular myomectomy saline injection in women undergoing laparoscopic myomectomy procedure
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — intracapsular injection of Terlipressin versus Carbetocin for decreasing blood loss in women undergoing laparoscopic myomectomy
  Other Names: carbitocin

SUMMARY:
Our study aims to evaluate the efficacy of intracapsular injection of Terlipressin versus Carbetocin injection on hemoglobin level in women undergoing abdominal laparoscopic myomectomy. Moreover, to evaluate their efficacy in decreasing blood loss on operative time and to describe the injection sequelae for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

DETAILED DESCRIPTION:
This study is a prospective, comparative, double-blinded randomized placebo-controlled trial and multi-center study that will be conducted at Wael ElBanna Clinic and the NRC site. The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants. Data will be pooled and presented in aggregate, without the identification of individual subjects. The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms:

* Arm 1: intramyometrial injection of Terlipressin in women undergoing laparoscopic myomectomy procedure
* Arm 2: intramyometrial injection of Carbetocin in women undergoing laparoscopic myomectomy procedure
* Arm 3: intramyometrial injection of saline in women undergoing laparoscopic myomectomy procedure Subjects who meet diagnostic requirements as listed in the inclusion and exclusion criteria will be included in the study. Women will be randomized to one of the three arms using a computer-generated randomization table with a 1:1:1 group allocation.

ELIGIBILITY:
Inclusion Criteria

1. Women aged 16-45 years
2. Appropriate medical status for laparoscopic surgery (largest myoma ≤15 cm)
3. Baseline hemoglobin ≥9 g/dl
4. No contra-indications to the use of glyopressin or carbitocin
5. Myoma-related symptoms, such as pelvic pressure or pain, menorrhagia, or infertility
6. Not pregnant at the time of presentation (i.e., negative urine pregnancy test or last menstrual period within the last 4 weeks)

Exclusion Criteria:

1. Previous myomectomy
2. History of bleeding disorders
3. Concurrent anticoagulation therapy
4. History of Uncontrolled ischaemic heart disease
5. Any pelvic abnormalities requiring concomitant surgery
6. Treatment with a GnRH agonist or ulipristal acetate within three months preceding surgery
7. Inability to understand and provide written informed consent

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women have multiple myomectomy undergoing laparoscopic myomectomy
Enrollment: 99 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
intracapsular injection of Terlipressin versus Carbetocin on change blood loss in patient in laparoscopic myomectomy | 12 hours
  measure the amount of blood loss in mm after intracapsular injection of Terlipressin versus Carbetocin versus saline as aplacebo in women undergoing laparoscopic myomectomy

SECONDARY OUTCOMES:
1. To evaluate the efficacy of intracapsular injection of Terlipressin versus Carbetocin on hemoglobin | 24 hours
  compare the hemoglobin level before and after operation after intracapsular injection of Terlipressin versus Carbetocin saline as aplacebo in women undergoing laparoscopic myomectomy
2. To evaluate the efficacy of intracapsular injection of Terlipressin versus Carbetocin on operative time | 12 hours
  2. To measure the operative time in minutes after intracapsular injection of Terlipressin versus Carbetocin versus saline as aplacebo in women undergoing laparoscopic myomectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Wael El Banna Clinic, Maadi, Egypt

REFERENCES:
- [Background] Marsh EE, Ekpo GE, Cardozo ER, Brocks M, Dune T, Cohen LS. Racial differences in fibroid prevalence and ultrasound findings in asymptomatic young women (18-30 years old): a pilot study. Fertil Steril. 2013 Jun;99(7):1951-7. doi: 10.1016/j.fertnstert.2013.02.017. Epub 2013 Mar 15. PMID 23498888
- [Background] Srivastava S, Mahey R, Kachhawa G, Bhatla N, Upadhyay AD, Kriplani A. Comparison of intramyometrial vasopressin plus rectal misoprostol with intramyometrial vasopressin alone to decrease blood loss during laparoscopic myomectomy: Randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:279-283. doi: 10.1016/j.ejogrb.2018.07.006. Epub 2018 Jul 5. PMID 30056355
- See also: Related Info — https://www.google.com/search?q=Srivastava+S%2C+Mahey+R%2C+Kachhawa+G%2C+Bhatla+N%2C+Upadhyay+AD%2C+Kriplani+A.+Comparison+of+intramyometrial+vasopressin+plus+rectal+misoprostol+with+intramyometrial+vasopressin+alone+to+decrease+blood+loss+during+laparoscopic+myomectomy%3A+Randomized+clinical+trial.+Eur+J+Obstet+Gynecol+Reprod+Biol.+2018+Sep%3B228%3A279%E2%80%9383.&oq=Srivastava+S%2C+Mahey+R%2C+Kachhawa+G%2C+Bhatla+N%2C+Upadhyay+AD%2C+Kriplani+A.+Comparison+of+intramyometrial+vasopressin+plus+rectal+misoprostol+with++intramyometrial+vasopressin+alone+to+decrease+blood+loss+during+laparoscopic+myomectomy%3A+Randomized+clinical+trial.+Eur+J+Obstet+Gynecol+Reprod+Biol.+2018+Sep%3B228%3A279%E2%80%9383.+&aqs=chrome..69i57.1122j0j15&sourceid=chrome&ie=UTF-8